CLINICAL TRIAL: NCT02337569
Title: A Randomized, Double-Blind, Placebo Controlled Study of NPC-02 in Patients With Zinc Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPC-02-4
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Zinc Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- NPC-02 (Experimental): Oral dose
  Interventions: Drug: NPC-02
- Placebo (Placebo Comparator): Oral dose
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: NPC-02
  Arms: NPC-02
Drug: Placebos
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate efficacy and safety of NPC-02 in patients with Zinc Deficiency.

ELIGIBILITY:
Inclusion Criteria:

The serum zinc concentrations are under the normal level before registration

Exclusion Criteria:

1. Heavy hepatitis
2. Malignant tumor
3. Severe heart disease, hematological disorder, kidney disease and pancreatic disease, etc.
4. The serum albumin under 2.8 g/dL
5. Patient of allergy and hyperesthesia to zinc containing medicine manufacturing (including supplement)
6. Patient who was taking a medicine including the zinc (including supplement) within 12 weeks before registration
7. Pregnant, suspected pregnant, lactating, patients who wish to have a child
8. Patient who participated in other clinical trials within 12 weeks before registration
9. Unsuitable as a target of this clinical trial judged by doctor

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The change amount of serum zinc concentration between starting and 8 weeks after dosing | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka, Japan

REFERENCES:
- [Derived] Katayama K, Hosui A, Sakai Y, Itou M, Matsuzaki Y, Takamori Y, Hosho K, Tsuru T, Takikawa Y, Michitaka K, Ogawa E, Miyoshi Y, Ito T, Ida S, Hamada I, Miyoshi K, Kodama H, Takehara T. Effects of Zinc Acetate on Serum Zinc Concentrations in Chronic Liver Diseases: a Multicenter, Double-Blind, Randomized, Placebo-Controlled Trial and a Dose Adjustment Trial. Biol Trace Elem Res. 2020 May;195(1):71-81. doi: 10.1007/s12011-019-01851-y. Epub 2019 Aug 7. PMID 31392541